CLINICAL TRIAL: NCT02125877
Title: A Randomized, Open-label, Multicenter, Two Arm, Phase II Study to Investigate the Benefits of an Improved Deferasirox Formulation (Film-coated Tablet)
Brief Title: Phase II Study to Investigate the Benefits of an Improved Deferasirox Formulation (Film-coated Tablet)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CICL670F2201
Record Dates: First submitted 2014-04-26; First posted 2014-04-29 (Estimated); Results first posted 2016-10-18 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Chronic Iron Overload Due to Transfusion-dependant Anemias
Keywords: Iron overload; Chelation; Thalassemia; Myelodysplastic syndrome (MDS); Transfusional hemisiderosis; Deferasirox; ICL670; Dispersible tablet; Film-coated tablet
MeSH Terms: conditions — Iron Overload; Thalassemia; Myelodysplastic Syndromes | interventions — Deferasirox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Deferasirox dispersible tablet (DFX-DT) (Active Comparator): Iron chelation naïve participants received DFX-DT 20 mg/kg/day once daily orally from weeks 1 - 4. After week 4, the dose could be adjusted by +/- 5 to 10 mg/kg/day, with a maximum dose of 40 mg/kg/day. Iron chelation pre-treated participants were supposed to start on a dose that was equivalent to their pre-washout dose.
  Interventions: Drug: Deferasirox dispersible tablet
- Deferasirox film-coated tablet (DFX-FCT) (Experimental): Participants received DFX-FCT 14 mg/kg/day once daily orally from weeks 1 - 4. After week 4, the dose could be adjusted by +/- 3.5 to 7 mg/kg/day, with a maximum dose of 28 mg/kg/day. Iron chelation pre-treated participants were supposed to start on a dose that was equivalent to their pre-washout dose
  Interventions: Drug: Defearisox film-coated tablet

INTERVENTIONS:
Drug: Deferasirox dispersible tablet — Deferasirox DT was provided as 125 mg, 250 mg and 500 mg dispersible tablets for oral use.
  Other Names: ICL670, DT (dispersible tablet)
  Arms: Deferasirox dispersible tablet (DFX-DT)
Drug: Defearisox film-coated tablet — Deferasirox FCT was provided as 90 mg, 180 mg and 360 mg film-coated tablets for oral use.
  Other Names: ICL670, FCT (film-coated tablet)
  Arms: Deferasirox film-coated tablet (DFX-FCT)

SUMMARY:
Assessed the new film-coated tablet formulation to the currently approved dispersible tablet formulation with regards to overall safety, Gastrointestinal (GI) tolerability, palatability, satisfaction and compliance

ELIGIBILITY:
Key Inclusion Criteria:

* Male and female patients aged ≥ 10 years
* Patients with transfusion-dependent thalassemia and iron overload, requiring deferasirox DT at doses of ≥ 30 mg/kg/day as per the investigator's decision OR Patients with very low, low or intermediate (int) risk myelodysplastic syndrome (MDS) and iron overload, requiring deferasirox DT at doses of ≥ 20 mg/kg/day as per the investigator's decision.
* History of transfusion of at least 20 PRBC units and anticipated to be transfused with at least 8 units of PRBCs annually during the study
* Serum ferritin > 1000 ng/mL, measured at screening Visit 1 and screening Visit 2 (the mean value will be used for eligibility criteria).

Key Exclusion Criteria:

* Creatinine clearance below the contraindication limit in the locally approved prescribing information. Creatinine clearance will be estimated from serum creatinine at screening Visit 1 and screening Visit 2 and the mean value will be used for eligibility criteria.
* Serum creatinine > 1.5 xULN at screening measured at screening Visit 1 and screening Visit 2 (the mean value will be used for eligibility criteria).
* ALT (SGPT) > 5xULN, unless LIC confirmed as >10 mg Fe/dw within 6 months prior to screening visit 1.
* Significant proteinuria as indicated by a urinary protein/creatinine ratio > 0.5 mg/mg in a non-first void urine sample at screening Visit 1 or screening Visit 2.
* Patients with significant impaired gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral deferasirox (e.g. ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
* Liver disease with severity of Child-Pugh Class B or C

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2014-07-08 (Actual); Primary Completion 2016-02-24 (Actual); Study Completion 2016-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (45):
- United States (5):
  - Children's Hospital of Orange County Onc Dept, Orange, California
  - Lurie Children's Hospital of Chicago Onc Dept, Chicago, Illinois
  - Children's Hospital Boston Department of Hematology, Boston, Massachusetts
  - Weill Cornell Medical College-Cornell University Onc Dept, New York, New York
  - Children's Hospital of Philadelphia Onc. Dept, Philadelphia, Pennsylvania
- Novartis Investigative Site, Buenos Aires, Argentina
- Austria (2):
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Vienna
- France (2):
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Paris
- Germany (7):
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Goslar
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Potsdam
- Greece (3):
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Patra - RIO, GR
  - Novartis Investigative Site, Thessaloniki, GR
- Italy (11):
  - Novartis Investigative Site, Brindisi, BR
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Cona, FE
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Cagliari, ITA
  - Novartis Investigative Site, Lecce, LE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Reggio Calabria, RC
  - Novartis Investigative Site, Verona, VR
  - Novartis Investigative Site, Napoli
- Novartis Investigative Site, Hazmiyeh, Beyrouth, Lebanon
- Malaysia (2):
  - Novartis Investigative Site, Kuala Lumpur
  - Novartis Investigative Site, Pulau Pinang
- Novartis Investigative Site, Mexico City, Mexico City, Mexico
- Novartis Investigative Site, Moscow, Russia, Russia
- Saudi Arabia (3):
  - Novartis Investigative Site, Dammam
  - Novartis Investigative Site, Jeddah
  - Novartis Investigative Site, Riyadh
- Spain (2):
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Bangkok, Thailand
- United Arab Emirates (2):
  - Novartis Investigative Site, Al Ain - Abu Dhabi, United Arab Emirates
  - Novartis Investigative Site, Dubai
- Novartis Investigative Site, London, United Kingdom

REFERENCES:
- [Derived] Taher AT, Origa R, Perrotta S, Kouraklis A, Ruffo GB, Kattamis A, Goh AS, Huang V, Zia A, Herranz RM, Porter JB. Patient-reported outcomes from a randomized phase II study of the deferasirox film-coated tablet in patients with transfusion-dependent anemias. Health Qual Life Outcomes. 2018 Nov 19;16(1):216. doi: 10.1186/s12955-018-1041-5. PMID 30453981

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized in a 1:1 ratio.
Period: Overall Study
Arm/Group | Deferasirox Dispersible Tablet (DFX-DT) | Deferasirox Film-coated Tablet (DFX-FCT)
Started | 86 | 87
Pharmacokinetic Analysis Set | 83 | 83
Pharmacokinetic Subset A | 16 | 15
Safety Set | 86 | 87
Completed | 73 | 77
Not Completed | 13 | 10
Not completed — Physician Decision | 1 | 0
Not completed — Death | 0 | 1
Not completed — Administrative problems | 0 | 1
Not completed — Participant/guardian decision | 0 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Protocol deviation | 4 | 1
Not completed — Adverse Event | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Deferasirox Dispersible Tablet (DFX-DT) | Deferasirox Film-coated Tablet (DFX-FCT) | Total
Number analyzed (Participants) | 86 | 87 | 173
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.1 (18.60) | 34.6 (19.97) | 34.9 (19.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 41 | 88
  Male | 39 | 46 | 85

OUTCOME MEASURES:

1. Primary Outcome: Overall Safety as Measured by Frequency of Adverse Events
Description: The percentage of participants with adverse events, serious adverse events and deaths was assessed.
Time Frame: 28 weeks
Population: The safety set, which included all participants who received at least one dose of study drug, was analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Deferasirox Dispersible Tablet (DFX-DT) | Deferasirox Film-coated Tablet (DFX-FCT)
Number analyzed (Participants) | 86 | 87
Percentage of participants
  Adverse events | 89.5 | 89.7
  SAEs | 15.1 | 18.4
  Deaths | 0 | 1.1

2. Primary Outcome: Overall Safety as Measured by Changes in Laboratory Values From Baseline
Description: The percentage of participants with post-baseline laboratory values meeting specified criteria for notable/extended range was assessed. The following laboratory parameters were measured: platelet count, absolute neutrophils, serum creatinine , creatinine clearance, urinary protein/urinary creatinine ratio, alanine aminotransferase (ALT) and aspartate aminotransferase (AST). Note that within data categories, creat = creatinine, cons = consecutive, ULN = upper limit of normal and urin = urinary.
Time Frame: baseline (BL), 30 weeks
Population: The safety set, which included all participants who received at least one dose of study drug, was analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Deferasirox Dispersible Tablet (DFX-DT) | Deferasirox Film-coated Tablet (DFX-FCT)
Number analyzed (Participants) | 86 | 87
Percentage of participants
  platelet count, notable range: <100 x 10^9/L | 9.3 | 8.0
  platelet count, extended range: <50 x 10^9/L | 3.5 | 5.7
  absolute neutrophils, notable range: <1.5 x 10^9/L | 8.1 | 13.8
  absolute neut., extended range: <0.5 x 10^9/L | 4.7 | 0
  serum creat, 2 cons >33% incr. from BL and >ULN | 4.7 | 3.4
  creat clearance, notable range: 2 cons <60mL/min | 7.0 | 2.3
  creat clearance, extended range: 2 cons <40mL/min | 2.3 | 2.3
  urin protein/urin creat ratio, 2 cons >1.0 mg/mg | 2.3 | 0
  ALT, notable range: >5 x ULN and >2 x BL | 1.2 | 1.1
  ALT, extended range: >10 x ULN and >2 x BL | 1.2 | 0
  AST, notable range: >5 x ULN and >2 x BL | 0 | 1.1
  AST, extended range: >10 x ULN and >2 x BL | 1.2 | 0

3. Secondary Outcome: Frequency of Selected Gastro-intestinal (GI) Adverse Events
Description: The percentage of participants with any GI adverse event, diarrhea, constipation, nausea, vomiting, abdominal pain was assessed.
Time Frame: 28 weeks
Population: The safety set, which included all participants who received at least one dose of study drug, was analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Deferasirox Dispersible Tablet (DFX-DT) | Deferasirox Film-coated Tablet (DFX-FCT)
Number analyzed (Participants) | 86 | 87
Percentage of participants
  Any GI adverse event | 61.6 | 58.6
  Abdominal pain | 26.7 | 26.4
  Constipation | 15.1 | 8.0
  Diarrhea | 34.9 | 33.3
  Nausea | 26.7 | 27.6
  Vomiting | 22.1 | 17.2

4. Secondary Outcome: Mean Domain Scores of the Modified Satisfaction With Iron Chelation Therapy (Modified SICT)
Description: The modified SICT consisted of 13 items that represent 3 domains: adherence, satisfaction and concerns. The adherence domain consisted of 7 items, 6 which were measured using a 5-point response scale and was calculated by summing the 6 items. The score range from 6 to 30 and higher scores indicated worse adherence. The satisfaction domain consisted of 3 items, 2 which were measured using a 5-point response scale and was calculated by summing the 2 items. The score range from 2 to 10 and higher scores indicated worse satisfaction. The concerns domain consisted of 3 items to address any concerns or worries with his/her medication. All 3 items were measured on a 5-point response scale and were calculated by summing the 3 items. The score range from 3 to 15 and higher scores indicated fewer concerns. For all three domains, the meaningful difference between two treatment arms was determined to be 1 point.
Time Frame: weeks 2, 3, 13 and 24 (end of treatment or within 7 days of last dose)
Population: The safety set, which included all participants who received at least one dose of study drug, was considered for the analysis. However, only participants with values at the given week were included in the analysis for that week.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Deferasirox Dispersible Tablet (DFX-DT) | Deferasirox Film-coated Tablet (DFX-FCT)
Number analyzed (Participants) | 86 | 87
score on a scale
  week 2, adherence (n=70,70) | 10.3 (3.80) | 7.6 (2.14)
  week 2, satisfaction/preference (n=70,70) | 5.2 (2.24) | 2.8 (1.37)
  week 2, concerns (n=70,70) | 12.9 (2.94) | 13.8 (2.02)
  week 3, adherence (n=58,51) | 10.9 (4.09) | 7.7 (2.06)
  week 3, satisfaction/preference (n=58,51) | 5.4 (2.22) | 2.6 (1.05)
  week 3, concerns (n=58,51) | 12.4 (2.73) | 14.0 (1.49)
  week 13, adherence (n=59,64) | 11.2 (3.56) | 7.8 (2.05)
  week 13, satisfaction/preference (n=59,64) | 5.4 (2.14) | 2.9 (1.54)
  week 13, concerns (n=59,64) | 12.7 (2.50) | 13.6 (1.87)
  week 24, adherence (n=63,60) | 12.5 (5.32) | 7.5 (2.41)
  week 24, satisfaction/preference (n=63,60) | 5.8 (2.28) | 2.9 (1.58)
  week 24, concerns (n=63,60) | 11.8 (3.07) | 13.7 (1.84)

5. Secondary Outcome: Palatability Questionnaire Score
Description: The palatability questionnaire consisted of 4 items. The first item measured the taste and aftertaste of the medication and were scored a on a 5-point response scale. The second item offered an additional response option of "no aftertaste". The last 2 items referred to whether the medication was taken, i.e. swallowed or vomited, and how the participant perceived the amount of medication to be taken. The palatability summary score was calculated using a scoring matrix from items 1, 3 and 4 scores and the score ranges from 0 - 11. Higher scores indicated the best palatability. A meaningful difference between two treatment arms was determined to be 1 point.
Time Frame: weeks 2, 3, 13 and 24 (end of treatment or within 7 days of last dose)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Deferasirox Dispersible Tablet (DFX-DT) | Deferasirox Film-coated Tablet (DFX-FCT)
Number analyzed (Participants) | 86 | 87
score on a scale
  week 2 (n=69,70) | 9.0 (3.01) | 10.8 (0.50)
  week 3 (n=57,51) | 8.8 (3.01) | 10.8 (0.45)
  week 13 (n=59,62) | 9.3 (2.84) | 10.8 (1.16)
  week 24 (n=63,60) | 8.8 (3.10) | 10.9 (0.34)

6. Secondary Outcome: Weekly Average of Daily Scores of the Gastrointestinal (GI) Symptom Diary
Description: The GI symptom diary consisted of 6 items, five which were scored using a 0 - 10 rating scale with item appropriate anchors to rate the symptom, for example, Pain in your belly: 0 = no pain and 10 = worst pain. The GI diary summary score was created using the 10 point response scale for the 5 items. The GI symptom daily diary had a minimum score of 0 and a maximum score of 50. The weekly average score for the 7 days was calculated for each individual item and the GI summary score was created from these weekly averages. Higher scores indicated worse symptoms. A meaningful difference between two treatment arms was determined to be 0.3 point.
Time Frame: weeks -1, 4, 8, 12, 16, 20, 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Deferasirox Dispersible Tablet (DFX-DT) | Deferasirox Film-coated Tablet (DFX-FCT)
Number analyzed (Participants) | 86 | 87
score on a scale
  week -1 (n=69,65) | 1.4 (2.10) | 1.9 (3.69)
  week 4 (n=60,64) | 1.8 (3.49) | 1.1 (2.15)
  week 8 (n=59,51) | 1.4 (2.45) | 1.1 (2.16)
  week 12 (n=51,45) | 1.7 (3.16) | 1.0 (1.78)
  week 16 (n=48,41) | 1.9 (3.75) | 0.9 (1.92)
  week 20 (n40,39) | 1.5 (3.27) | 0.9 (1.44)
  week 24 (n32,26) | 1.5 (3.29) | 1.2 (1.89)

7. Secondary Outcome: Number of Participants With Weekly Average Compliance of Medication Consumption
Description: A compliance questionnaire assessed whether the medication was taken. Weekly average compliance was calculated when there were at least four non-missing daily responses.
Time Frame: Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24
Population: The safety set, which included all participants who received at least one dose of study drug, was analyzed.
Measure: Number; unit: Participants
Arm/Group | Deferasirox Dispersible Tablet (DFX-DT) | Deferasirox Film-coated Tablet (DFX-FCT)
Number analyzed (Participants) | 86 | 87
Participants
  week 1 | 56 | 53
  week 2 | 64 | 64
  week 3 | 62 | 56
  week 4 | 58 | 58
  week 5 | 56 | 58
  week 6 | 62 | 51
  week 7 | 55 | 48
  week 8 | 56 | 46
  week 9 | 53 | 45
  week 10 | 52 | 46
  week 11 | 50 | 42
  week 12 | 50 | 41
  week 13 | 49 | 47
  week 14 | 51 | 42
  week 15 | 48 | 42
  week 16 | 48 | 40
  week 17 | 43 | 39
  week 18 | 43 | 38
  week 19 | 40 | 37
  week 20 | 40 | 36
  week 21 | 39 | 36
  week 22 | 38 | 34
  week 23 | 36 | 33
  week 24 | 30 | 24

8. Secondary Outcome: Weekly Dose Violation Rate
Description: The dose violation is defined as a dose either missed completely or not taken in accordance with the timing instruction (no later than 12:00 pm. The rate was calculated as [number of dose violations/drug exposure (days)] x 100.
Time Frame: weeks 1, 4, 8, 12, 16, 20, 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent dose violation
Arm/Group | Deferasirox Dispersible Tablet (DFX-DT) | Deferasirox Film-coated Tablet (DFX-FCT)
Number analyzed (Participants) | 86 | 87
percent dose violation
  week 1 (n=56,53) | 17.7 (31.04) | 15.8 (29.42)
  week 4 (n=58,58) | 15.8 (32.51) | 6.7 (15.45)
  week 8 (n=56,46) | 18.0 (35.38) | 8.4 (22.17)
  week 12 (n=50,41) | 15.7 (34.22) | 10.7 (22.63)
  week 16 (n=48,40) | 13.5 (31.08) | 10.0 (24.5)
  week 20 (n=40,36) | 22.6 (38.38) | 11.3 (26.67)
  week 24 (n=30,24) | 17.1 (34.26) | 10.1 (25.47)

9. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Quantifiable Concentration (AUClast)
Description: Blood samples were collected to assess AUClast.
Time Frame: week 1, day 1: pre-dose (0 hour) and 1, 2, 3, 4, 8 and 24 hours post dose; week 3, day 1: pre-dose (0 hour) and 1, 2, 3, 4, 8 and 24 hours post dose
Population: The Pharmacokinetic subset A analysis set was considered for the analysis, but only participants with non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: umol/L*h
Arm/Group | Deferasirox Dispersible Tablet (DFX-DT) | Deferasirox Film-coated Tablet (DFX-FCT)
Number analyzed (Participants) | 16 | 15
umol/L*h
  week1 (n=14,15) | 1110 (495) | 1040 (405)
  week 3 (n=13,15) | 1590 (540) | 2110 (987)

10. Secondary Outcome: Observed Maximum Plasma Concentration Following Drug Administration (Cmax)
Description: Blood samples were collected to assess Cmax.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Deferasirox Dispersible Tablet (DFX-DT) | Deferasirox Film-coated Tablet (DFX-FCT)
Number analyzed (Participants) | 16 | 15
umol/L
  week 1 (n=14,15) | 74.6 (30.7) | 79.3 (23.5)
  week 3 (n=14,15) | 118 (82.3) | 139 (57.2)

11. Secondary Outcome: Time to Reach the Maximum Plasma Concentration After Drug Administration (Tmax)
Description: Blood samples were collected to assess Tmax.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Median (Full Range); unit: hour
Arm/Group | Deferasirox Dispersible Tablet (DFX-DT) | Deferasirox Film-coated Tablet (DFX-FCT)
Number analyzed (Participants) | 16 | 15
hour
  week 1 (n=14,15) | 3.57 [1.15 to 7.89] | 2.00 [1.15 to 15.6]
  week 3 (n=14,15) | 2.85 [1.40 to 8.39] | 2.02 [1.07 to 5.06]

12. Secondary Outcome: Dererasirox Plasma Concentration
Description: Blood samples were collected to assess deferasirox concentration. Dose-adjusted calculations are presented: (concentration/actual dose)*20 for participants on DFX-DT and (concentration/actual dose)*14 for participants on DFX-FCT.
Time Frame: Week 3, day 1, pre-dose (0 hour (h)) and 2 h post-dose; week 13, day 1, pre-dose (0 hour (h)) and 2 h post-dose; and week 21, day 1, pre-dose (0 hour (h)) and 2 h post-dose
Population: The Pharmacokinetic analysis set for all participants was considered for this analysis, but only participants with non-missing values were included in the analysis.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Deferasirox Dispersible Tablet (DFX-DT) | Deferasirox Film-coated Tablet (DFX-FCT)
Number analyzed (Participants) | 83 | 83
umol/L
  week 3, pre-dose (n=63,70) | 39.6 (48.4) | 27.3 (20.4)
  week 3, 2 hours post-dose (n=67,76) | 80.8 (52.2) | 95.5 (53.0)
  week 13, pre-dose (n=69.56) | 37.1 (37.8) | 31.3 (22.9)
  week 13, 2 hours post-dose (n=74,59) | 78.7 (39.5) | 92.5 (39.1)
  week 21, pre-dose (n=54,59) | 46.6 (46.4) | 43.1 (36.8)
  week 21, 2 hours post-dose (n=59,64) | 89.8 (59.3) | 105 (51.2)

ADVERSE EVENTS:
Arm/Group | Deferasirox Dispersible Tablet (DFX-DT) | Deferasirox Film-coated Tablet (DFX-FCT)
Serious Adverse Events (participants affected / at risk) | 13/86 | 16/87
Other Adverse Events (participants affected / at risk) | 69/86 | 72/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Deferasirox Dispersible Tablet (DFX-DT) (N=86) | Deferasirox Film-coated Tablet (DFX-FCT) (N=87)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Haemolysis (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 0
Neutropenic colitis (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Face oedema (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Brucellosis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Post procedural pneumonia (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 2
Septic shock (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 2
Delayed haemolytic transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Ejection fraction decreased (Investigations) | 1 | 0
Urine protein/creatinine ratio increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Deferasirox Dispersible Tablet (DFX-DT) (N=86) | Deferasirox Film-coated Tablet (DFX-FCT) (N=87)
Abdominal pain (Gastrointestinal disorders) | 23 | 23
Abdominal pain upper (Gastrointestinal disorders) | 6 | 10
Constipation (Gastrointestinal disorders) | 13 | 7
Diarrhoea (Gastrointestinal disorders) | 30 | 27
Dyspepsia (Gastrointestinal disorders) | 2 | 6
Nausea (Gastrointestinal disorders) | 23 | 24
Vomiting (Gastrointestinal disorders) | 18 | 15
Asthenia (General disorders) | 8 | 4
Fatigue (General disorders) | 7 | 5
Pyrexia (General disorders) | 7 | 7
Bacteriuria (Infections and infestations) | 5 | 5
Gastroenteritis (Infections and infestations) | 3 | 5
Influenza (Infections and infestations) | 5 | 0
Upper respiratory tract infection (Infections and infestations) | 6 | 6
Urinary tract infection (Infections and infestations) | 6 | 3
Blood creatinine increased (Investigations) | 7 | 8
Urine protein/creatinine ratio increased (Investigations) | 11 | 17
Hyperphosphataemia (Metabolism and nutrition disorders) | 5 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 4
Headache (Nervous system disorders) | 12 | 5
Haematuria (Renal and urinary disorders) | 2 | 8
Proteinuria (Renal and urinary disorders) | 4 | 8
Pyuria (Renal and urinary disorders) | 2 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.